CLINICAL TRIAL: NCT04674137
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Pilot Study to Assess the Efficacy and Safety of XC8 in Patients With the Eosinophilic Phenotype of Bronchial Asthma
Brief Title: XC8 in the Treatment of Patients With the Eosinophilic Phenotype of Bronchial Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chemlmmune Therapeutics LLC (Industry)
Collaborators: EURRUS Biotech GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PULM-XC8-04
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Bronchial Asthma; Eosinophilic Asthma
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia | interventions — histamine glutarimide

STUDY DESIGN:
Intervention Model Description: At Visit 3, Week 0 all patients were randomized into 2 groups in 1:1 ratio (35 patients to group of XC8 100 mg and 35 patients to Placebo group).
Who Masked: Participant, Investigator
Masking Description: For blinding purposes the Placebo was made with the corresponding labelling of the study drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XC8 100 mg (Experimental): XC8 100 mg orally
  Interventions: Drug: XC8 100 mg
- Placebo (Placebo Comparator): Placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XC8 100 mg — 1 tablet of XC8 100 mg once daily in the morning during 12 weeks of treatment period.
  Other Names: Histamine glutarimide
  Arms: XC8 100 mg
Drug: Placebo — 1 tablet of placebo once daily in the morning during 12 weeks of treatment period.
  Arms: Placebo

SUMMARY:
A multicenter, double-blind, randomized, pilot study in parallel groups to assess the efficacy and safety of XC8 at a dose of 100 mg versus placebo over a 12-week treatment period in non-smoking patients with a confirmed bronchial asthma (BA) and the eosinophil blood level 2 times within 1 week interval of ≥ 300 cells/μl.

Study design was developed by Chemlmmune Therapeutics LLC, Russia in cooperation with Eurrus Biotech GmbH, Austria.

DETAILED DESCRIPTION:
The study consists of 3 periods: screening (2 weeks), treatment period (12 weeks) and follow-up (2 weeks). All eligible patients are randomized into one of two treatment groups in a ratio of 1:1. During the study patients will continue to receive stable doses of inhaled corticosteroids (ICS) with or without the long-acting β2-agonists; when required, patients will receive short-acting β2-agonists.The randomized patients will be stratified by the site, baseline forced expiratory volume (FEV1) in the range of 55 to 70% and 71% to 85%, and therapy of BA (inhaled corticosteroids (ICS) with or without long-acting β2 agonists).

The Study drug is produced by Hennig Arzneimittel GmbH und Co., Germany.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form;
2. Male and female non-smokers of 18 to 65 years of age (inclusive);
3. The diagnosis of asthma not earlier than 12 months prior to screening;
4. Steps 2 and 3 according to Global Initiative for Asthma (GINA, 2019) recommendations;
5. Patients receiving stable ICS doses with or without long-acting β2-agonists;
6. Еosinophil blood level measured twice at a 1 week interval, of ≥ 300 cells/µl ;
7. Signs of partially controlled BA within 4 weeks prior to screening according to GINA 2019 recommendations;
8. FEV1 value prior to the use of bronchodilators in the range of 55 to 85% of the proper value (inclusive);
9. Consent of patients to use adequate contraception methods throughout the study;
10. Ability to comply with all the study protocol requirements.

Exclusion Criteria:

1. Pregnant or lactating women, or women planning to get pregnant during the clinical study; women of child-bearing potential (including those without history of surgical sterilization and women with <2 years post-menopause) not using adequate contraception methods;
2. Smoking for 1 year prior to screening or previous smoking history of more than 10 packs/year;
3. Severe exacerbations or uncontrolled BA within 3 months prior to screening;
4. Chronic obstructive pulmonary disease (COPD) or other serious lung diseases other than asthma;
5. Inflammatory diseases of the oral cavity at screening;
6. An acute infectious disease within 30 days prior to screening;
7. Participation in any clinical study or any study drug administration within 30 days prior to screening;
8. Taking or indications for taking of prohibited drugs (including anti-leukotriene preparations, modified-release theophylline, etc.);
9. Indications for long-term use of systemic steroids or nonsteroidal anti-inflammatory drugs or drugs affecting on the immune system;
10. The need for periodical intake of antihistamines during the study (stable doses of antihistamines for at least 1 month prior to screening and throughout the study is allowed);
11. Immunosuppressant therapy within 3 months prior to screening;
12. Anaphylaxis, generalized urticaria, or angioedema within 1 year prior to screening;
13. Known allergies, hypersensitivity or contraindications for XC8 or its ingredients;
14. A history of systemic autoimmune diseases or vascular collagenosis;
15. Malignancies within the last 5 years (except for the cured basal cell carcinoma);
16. Significant cardiovascular diseases diagnosed at present or within 12 months prior to screening; uncontrolled hypertension with systolic blood pressure > 180 mm Hg and diastolic blood pressure > 110 mm Hg; pulmonary embolism or deep vein thrombosis;
17. Nephrotic syndrome, moderate to severe chronic renal failure or significant renal impairment with creatinine level >1.5 mg/dL (132 μM/l) in males and > 1.4 mg/dL (123 μM/l) in females or glomerular filtration rate < 60 mL/min;
18. HIV, hepatitis B or C, history of cirrhosis; 3-fold increased serum aspartate aminotransferase or alanine aminotransferase > above the Upper Limit of Normal; 2-fold increased total bilirubin level > above at screening;
19. Anemia (hemoglobin level ≤ 10.5 g/dL in females or ≤ 11.5 g/dL in males); significant blood loss or collection of at least one volumetric unit of donated blood (> 500 mL), or blood transfusion within 12 weeks prior to screening;
20. Any concomitant disease, other than asthma, not controlled by a stable therapy regimen;
21. Drugs or alcohol abuse at screening or in the past, which, in the Investigator's opinion, makes the patient not eligible for participation in the study;
22. Inability to read or write; unwillingness to understand and comply with the protocol procedures; non-compliance with the drug dosing regimen or procedures which, in the Investigator's opinion, may affect study results or the patient's safety and prevent the patient's participation in the study; any other concomitant diseases or severe mental disorders, which make the patient ineligible for participation in the study, limit the legal basis for Informed Consent procedure, or may affect the patient's ability to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Rate of achieving the minimal clinically significant absolute change in FEV1 (+200 mL) | Week 0 - Week 12
  To assess the rate of achieving minimal clinically significant absolute change in FEV1 measured in mL compared to baseline through spirometry testing.

SECONDARY OUTCOMES:
Changes in FEV1 (in mL) | Week 0 - Week 12
  To assess relative and absolute changes in FEV1 prior to the use of bronchodilators (in mL)
Changes in FEV1 (in % of predicted) | Week 0 - Week 12
  To assess relative and absolute changes in FEV1 prior to the use of bronchodilators (in % of predicted value)
Change in Peak Expiratory Flow (PEF) Rate | Week 0 - Week 12
  To assess daily variability of PEF rate measured in the morning and evening
Change in forced vital capacity of lungs (FVC) in % of predicted | Week 0 - Week 12
  To assess changes in FVC measured through spirometry testing
Change in FEV1/FVC (in % of predicted) | Week 0 - Week 12
  To assess changes in FEV1/FVC measured through spirometry testing
Change in forced expiratory flow (FEF) 25-75% (in % of predicted) | Week 0 - Week 12
  To assess changes in FEF 25-75% measured through spirometry testing
Rate of exacerbations of BA | Week 0 - Week 12
  To assess the number of patients with exacerbations of BA by GINA 2019 Criteria
Change in the Asthma Control Questionnaire 7 (ACQ-7) scores | Week 0 - Week 12
  To assess the changes in ACQ-7
Number of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Week 0 - Week 14
  AEs will be summarized descriptively by treatment arm. Verbatim terms will be mapped to preferred terms and organ systems using the current Medical Dictionary for Regulatory Activities (medDRA).

CONTACTS AND LOCATIONS:
Locations (18):
- Russia (18):
  - Federal State Autonomous Educational Institution of Higher Education "Immanuel Kant Baltic Federal University"of Ministry of Health of the Russian Federation, Kaliningrad
  - Federal State Autonomous Educational Institution of Higher Education "Kazan (Volga region) Federal University", Kazan'
  - Federal State Educational Institution of Higher Education "Kazan State Medical University" of the Ministry of Health of the Russian Federation, Kazan'
  - State Budgetary Institution of Healthcare of Moscow "City Clinical Hospital n.a. D.D.Pletnev" of the Moscow Department of Healthcare", Moscow
  - State Budgetary Institution of Healthcare of Moscow "City Clinical Hospital No. 52" of the Moscow Department of Healthcare, Moscow
  - Federal State Educational Institution of Higher Education "Moscow State University of Medicine and Dentistry n.a.A.I.Yevdokimov" of Ministry of Health of the Russian Federation, Moscow
  - State Budgetary Health Institution Republic of Karelia "Republican Hospital named V.A.Baranov", Petrozavodsk
  - JSC "Polyclinic complex", Saint Petersburg
  - State Budgetary Institution of Healthcare "Leningrad region Clinical Hospital", Saint Petersburg
  - LLC "Medical Center" Reavita Med St. Petersburg", Saint Petersburg
  - Saint Petersburg State Budgetary Institution of Healthcare "City polyclinic №117", Saint Petersburg
  - Saint Petersburg State Budgetary Institution of Healthcare St. Martyr Elizabeth City Hospital", Saint Petersburg
  - LLS Research Center for Eco-Security, Saint Petersburg
  - Federal State Autonomous Educational Institution of Higher Education "Pavlov First Saint Petersburg State Medical University"of the Ministry of Health of the Russian Federation, Saint Petersburg
  - LLS "Mayle", Saint Petersburg
  - State Healthcare Institution "Regional Clinical Hospital", Saratov
  - LLS diagnostic clinic "Konstanta", Yaroslavl
  - State autonomous healthcare institution of Yaroslavl Region "Сlinical hospital for emergency medical care n. a. N.V. Solovyov" of Ministry of Health of the Russian Federation, Yaroslavl

IPD SHARING:
Plan to Share IPD: No